CLINICAL TRIAL: NCT01969149
Title: Intravenous Exenatide (Byetta®) Versus Insulin for Perioperative Glycemic Control in Cardiac Surgery: the Open-labeled Randomized Phase II/III ExStress Study
Brief Title: Exenatide for Stress Hyperglycemia
Acronym: ExSTRESS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: AstraZeneca (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: API/2009/10
Record Dates: First submitted 2013-10-15; First posted 2013-10-25 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2016-03

CONDITIONS: Stress Hyperglycemia
Keywords: Stress Hyperglycemia; Perioperative glycemic control; Cardiac surgery; Coronary artery bypass surgery
MeSH Terms: interventions — Exenatide; Incretins; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide group (Experimental): Exenatide. Exenatide: bolus of 0.05 µg/min infused during the 1st hour of treatment, followed by a continuous infusion of 0.025 µg/min until the end of treatment.
  The exenatide therapy will begin as soon as a blood glucose level is above 140 mg/dl will be measured. A of exenatide will be intravenously .
  The treatment will be administrated during the first postoperative 48 hours in the intensive care unit or until intensive care unit discharge if this event occurs earlier.
  Interventions: Drug: Exenatide
- Insulin group (Active Comparator): Insulin: Humalog (insulin lispro human analog). The insulin therapy will begin as soon as a blood glucose level is above 140 mg/dl will be measured.
  The dose of insulin intravenously infused will be adapted to blood glucose measurements, following the insulin therapy protocol used in our department.
  The insulin therapy protocol used in our department and prescribed as the benchmark treatment in the present study has been validated in a previous study. It has been derived from the protocol validated by Goldberg et al.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Exenatide
  Other Names: Byetta; Exendin-4; Incretin
  Arms: Exenatide group
Drug: Insulin
  Other Names: Humalog Insulin Lispro Human Analog
  Arms: Insulin group

SUMMARY:
Stress hyperglycemia is a common phenomenon in cardiac surgery that concerns diabetic and non diabetic patients.

It has been shown that perioperative hyperglycemia is an independent risk factor of postoperative mortality and morbidity.

The Leuven et al.'s study suggested that strict glycemic perioperative control using an intensive insulin therapy could reduce mortality and morbidity in surgical intensive care's patients. This study included a majority of cardiac surgery patients. Others studies have suggested that the beneficial effect of insulin-based tight perioperative glycemic control might be hampered by iatrogenic hypoglycemia. Moreover, insulin therapy failed to obtain perioperative glycemic stability in most patients.

Exenatide (Byetta ®) is an incretin mimetic, characterized by an anti-hyperglycemic effect that depends on the blood glucose level.

We hypothesize that continuous intravenous infusion of exenatide could improve perioperative glycemic control and stability and could reduce the risk of iatrogenic hypoglycemia compared to a conventional insulin therapy during the perioperative period of cardiac surgery.

DETAILED DESCRIPTION:
The phase II of the study will assess the safety and the efficacy of a continuous intravenous infusion of exenatide for the management of post operative stress hyperglycemia after planned coronary artery graft bypass (CABG) surgery.

A nested cohort study will concern the 24 first patients included in the study (12 patients/group) to assess the impact of a continuous intravenous infusion of exenatide on post operative glycemic variability after planned CABG surgery.

The aim of the phase III of the study will compare the efficacy of a continuous intravenous infusion of exenatide to the gold standard treatment, i.e the intravenous infusion of short-acting insulin, for the management of post operative stress hyperglycemia after planned CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18.
* Patient consent.
* Non insulin requiring type 2 diabetic patients.
* Non diabetic patients.
* Planned coronary artery bypass graft (CABG) surgery.
* ASA (American Society of Anesthesiologists) score 1, 2, or 3.

Exclusion Criteria:

* Pregnancy and breast feeding.
* Pancreatectomy.
* Acute pancreatitis.
* Chronic pancreatitis.
* Type 1 diabetic patients.
* Insulin requiring type 2 patients.
* HbA1c>8%
* Ketoacidosis.
* Hyperosmolar coma.
* Preoperative blood glucose level above 300 mg/dl [21].
* Insulin or exenatide contraindication.
* History of renal transplantation or currently receiving renal dialysis or creatinine clearance below 60 ml/min.
* Emergency surgery.
* Planned non CABG cardiac surgery.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients spending more than 50 % of the time in the glycemic target range (100 to 140 mg/dl) | 48 hours
  The percentage of time spent achieving blood glucose control is defined as the ratio between the total time spent achieving blood glucose control and the total time under treatment.
  Blood glucose measurement will be done hourly. Blood glucose control is considered to be achieved between 2 blood glucose measurements if the first blood glucose value measured belongs to blood glucose target interval, defined as blood glucose level between 100 mg/dl l and 140 mg/dl l.

SECONDARY OUTCOMES:
Hypoglycemia | 48 hours
  Hypoglycemia is defined as blood glucose level less than 80 mg/dl.
Severe hypoglycemia | 48 hours
  Severe hypoglycemia is defined as blood glucose level less than 40 mg/dl.
Number of patients needing rescue to insulin therapy protocol | 48 hours
Number of adverse events occuring in the exenatide group | Day 30
  As the safety of exenatide has never been assessed in the perioperative period in cardiac surgery, all adverse events will be reported, in particular: known adverse events (diarrhea, nausea, vomiting) et severe adverse events (pancreatitis, acute renal failure, death, cardiac arrest).
Mortality | Day 30
Postoperative morbidity | Day 30
  Postoperative morbidity is defined as:
  * neurological complications: stroke.
  * renal complication: acute renal failure requiring dialysis.
  * cardiac complication: cardiogenic shock, arrhythmia, myocardial infarct.
  * vasopressive drug support in postoperative intensive care unit.
  * length of postoperative mechanical ventilation.
  * infectious complication: deep sternal infection.
The mean (GluAve) and standard deviation (GluSD) of blood glucose | 48 hours
The coefficient of variability (GluCV) of blood glucose level | 48 hours
  GluCV = GluSD*100/GluAve
Mean number of blood glucose measured | 48 hours
Mean difference between each blood glucose measurement and 120 mg/dl | 48 hours
Perioperative cardiac mortality | Day 30
Perioperative non cardiac mortality | Day 30
Length of stay in intensive care unit | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Besch, MD, Principal Investigator — CHRU Besançon; Sébastien Pili-Floury, MD, PhD, Study Director — CHRU Besançon
Locations (1):
- Post operative intensive care unit of the cardiac surgery department, Besançon, France

REFERENCES:
- [Background] Goldberg PA, Sakharova OV, Barrett PW, Falko LN, Roussel MG, Bak L, Blake-Holmes D, Marieb NJ, Inzucchi SE. Improving glycemic control in the cardiothoracic intensive care unit: clinical experience in two hospital settings. J Cardiothorac Vasc Anesth. 2004 Dec;18(6):690-7. doi: 10.1053/j.jvca.2004.08.003. PMID 15650975
- [Background] Studer C, Sankou W, Penfornis A, Pili-Floury S, Puyraveau M, Cordier A, Etievent JP, Samain E. Efficacy and safety of an insulin infusion protocol during and after cardiac surgery. Diabetes Metab. 2010 Feb;36(1):71-8. doi: 10.1016/j.diabet.2009.05.008. Epub 2010 Jan 25. PMID 20097589
- [Background] Galiatsatos P, Gibson BR, Rabiee A, Carlson O, Egan JM, Shannon RP, Andersen DK, Elahi D. The glucoregulatory benefits of glucagon-like peptide-1 (7-36) amide infusion during intensive insulin therapy in critically ill surgical patients: a pilot study. Crit Care Med. 2014 Mar;42(3):638-45. doi: 10.1097/CCM.0000000000000035. PMID 24247476
- [Derived] Besch G, Perrotti A, Salomon du Mont L, Puyraveau M, Ben-Said X, Baltres M, Barrucand B, Flicoteaux G, Vettoretti L, Samain E, Chocron S, Pili-Floury S. Impact of intravenous exenatide infusion for perioperative blood glucose control on myocardial ischemia-reperfusion injuries after coronary artery bypass graft surgery: sub study of the phase II/III ExSTRESS randomized trial. Cardiovasc Diabetol. 2018 Nov 1;17(1):140. doi: 10.1186/s12933-018-0784-y. PMID 30384842